CLINICAL TRIAL: NCT00871000
Title: Immunogenicity and Safety of GSK Biologicals' dTpa-IPV Vaccine (Boostrix Polio) as a Booster Dose in 5 to 6-year-old Children.
Brief Title: Immunogenicity and Safety of Boostrix Polio Vaccine as a Booster Dose in 5 to 6-year-old Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111815
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria; Poliomyelitis
Keywords: Boostrix Polio; dTpa-IPV
MeSH Terms: conditions — Tetanus; Diphtheria; Poliomyelitis | interventions — DTPa-HBV-IPV combined vaccine

ARMS (2):
- BOOSTRIX POLIO GROUP (Experimental): Healthy male or female children, between and including 5 to 6 years of age, who were primed with three doses of Infanrix™ vaccine according to the Italian 3-5-11 month vaccination schedule, additionally received a single booster dose of Boostrix Polio™ vaccine co-administered with a single dose of Priorix Tetra™ vaccine at Day 0. Boostrix Polio™ vaccine was administered intramuscularly in the deltoid region of the left upper arm, while the Priorix Tetra™ vaccine was administered subcutaneously in the deltoid region of the right upper arm.
  Interventions: Biological: Boostrix Polio™ 711866; Biological: Priorix Tetra TM 208136
- TETRAVAC GROUP (Active Comparator): Healthy male or female children, between and including 5 to 6 years of age, who were primed with three doses of Infanrix™ vaccine according to the Italian 3-5-11 month vaccination schedule, additionally received a single booster dose of Tetravac™ vaccine co-administered with a single dose of Priorix Tetra™ vaccine at Day 0. Tetravac™ vaccine was administered intramuscularly in the deltoid region of the left upper arm, while the Priorix Tetra™ vaccine was administered subcutaneously in the deltoid region of the right upper arm.
  Interventions: Biological: Priorix Tetra TM 208136; Biological: Tetravac TM

INTERVENTIONS:
Biological: Boostrix Polio™ 711866 — Single dose, intramuscular administration.
  Other Names: dTpa-IPV
  Arms: BOOSTRIX POLIO GROUP
Biological: Priorix Tetra TM 208136 — Single dose, subcutaneously.
  Other Names: MMRV
Biological: Tetravac TM — Single dose, intramuscular administration.
  Other Names: DTPa-IPV
  Arms: TETRAVAC GROUP

SUMMARY:
This phase 3b study will compare the immunogenicity and reactogenicity of the dTpa-IPV vaccine to that of a DTPa-IPV vaccine when administered as a booster dose in healthy children 5-6 years of age who have received three primary vaccination doses of DTPa-based vaccine according to the "3-5-11" month schedule recommended in Italy.

In this study, MMRV vaccine will also be co-administered to all children.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child of 5 and 6 years of age at the time of vaccination.
* Subjects who received a complete 3-dose vaccination with a DTPa-based combined vaccine according to a 3-5-11 month schedule in line with recommendations in Italy.
* Subjects who received a first dose of a live attenuated measles-mumps-rubella vaccine in the second year of life, in line with recommendations in Italy.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccine dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous booster vaccination against tetanus, diphtheria, pertussis and/or poliomyelitis since vaccination in the first two years of life.
* Previous measles, mumps, rubella and/or varicella second dose vaccination.
* Known history of diphtheria, tetanus, pertussis, poliomyelitis, measles, mumps, rubella and/or varicella disease.
* Known exposure to measles, mumps, rubella and/or varicella within 30 days prior to study start.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulin and/or any blood products within the three months preceding vaccination or planned administration during the study period.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Occurrence of any of the following adverse events after a previous administration of a DTP vaccine:

  * Hypersensitivity reaction to any component of the vaccine;
  * Encephalopathy of unknown aetiology occurring within 7 days following previous vaccination with pertussis-containing vaccine;
  * Fever >= 40°C within 48 hours of vaccination, not due to another identifiable cause;
  * Collapse or shock-like state within 48 hours of vaccination;
  * Convulsions with or without fever, occurring within 3 days of vaccination.
* Residence in the same household as a person high risk for varicella
* The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met:

  * Current febrile illness or axillary temperature ≥ 38.5 ºC or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2009-04-01; Primary Completion 2009-11-18 (Actual); Study Completion 2009-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Italy (8):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Modica (RG), Sicily
  - GSK Investigational Site, Ragusa, Sicily
  - GSK Investigational Site, Vittoria (RG)

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ferrera G, Cuccia M, Mereu G, Icardi G, Bona G, Esposito S, Marchetti F, Messier M, Kuriyakose S, Hardt K. Booster vaccination of pre-school children with reduced-antigen-content diphtheria-tetanus-acellular pertussis-inactivated poliovirus vaccine co-administered with measles-mumps-rubella-varicella vaccine: a randomized, controlled trial in children primed according to a 2 + 1 schedule in infancy. Hum Vaccin Immunother. 2012 Mar;8(3):355-62. doi: 10.4161/hv.18650. Epub 2012 Feb 13. PMID 22327497
- [Background] Ferrera G et al. A comparison of the immunogenicity and safety of a booster dose of reduced-antigen-content with full-strength DTPa-IPV vaccines administered with MMRV to children 5-6 years of age. Abstract presented at the 44th Congresso Nazionale Societa Italiana di Igiene, Medicina Preventiva e Sanita Pubblica (SITI). Venezia, Italia, 3-6 October, 2010.
- [Background] Ferrera G et al. Immunogenicity and safety of Booster vaccination with reduced-antigen-content or full-strength Diphtheria-Tetanus-Acellular-Pertussis-IPV vaccines in pre-school children, primed with a 2+1 schedule. Abstract presented at the 29th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID). The Hague, The Netherlands, 7-11 June 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 111815 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111815 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111815 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111815 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111815 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111815 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111815 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Boostrix Polio Group | Tetravac Group
Started | 151 | 152
Completed | 150 | 152
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix Polio Group | Tetravac Group | Total
Number analyzed (Participants) | 151 | 152 | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5 (0.14) | 5 (0.14) | 5 (0.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 68 | 149
  Male | 70 | 84 | 154
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 1 | 0 | 1
  Asian-Central/South Asian heritage | 1 | 4 | 5
  White-Arabic/North African heritage | 2 | 0 | 2
  White-Caucasian/European heritage | 147 | 147 | 294
  Not specified | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL). The reference cut-off value was greater than or equal to (≥) 0.1 IU/mL.
Time Frame: At Month 1, one month post-vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who had received the booster dose of study/comparator vaccine and for whom immunogenicity data and assay results for antibodies against at least one study vaccine antigen component were available.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 144
IU/mL
  Anti-D | 9.207 [8.057 to 10.522] | 21.393 [19.165 to 23.88]
  Anti-T | 12.527 [10.957 to 14.323] | 11.07 [9.872 to 12.413]

2. Primary Outcome: Anti-poliovirus Types 1, 2 and 3 Antibody Titres
Description: Antibody titers were presented as geometric mean titers (GMTs) for the assay cut-off ≥ the value of 8.
Time Frame: At Month 1, one month post-vaccination
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who had received the booster dose of study/comparator vaccine and for whom immunogenicity data and assay results for antibodies against at least one study vaccine antigen component were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 144
Titers
  Anti-Polio 1 | 1145.6 [978.7 to 1340.9] | 948 [817.5 to 1099.4]
  Anti-Polio 2 | 1076.4 [908.7 to 1274.9] | 1315.3 [1123.1 to 1540.3]
  Anti-Polio 3: number analyzed (Participants) | 138 | 144
  Anti-Polio 3 | 1937.8 [1631.4 to 2301.8] | 1657.3 [1385.5 to 1982.6]

3. Primary Outcome: Number of Seroprotected Subjects Against Polio Types 1, 2 and 3
Description: A seroprotected subject was defined as a subject with anti-polio types 1, 2 and 3 titers ≥ the value of 8. Antibody titers have been assessed by neutralization assay.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 144
Participants
  Anti-Polio 1 | 139 | 144
  Anti-Polio 2 | 139 | 144
  Anti-Polio 3: number analyzed (Participants) | 138 | 144
  Anti-Polio 3 | 138 | 144
Statistical Analysis 1: Comparison: Boostrix Polio Group vs Tetravac Group; To demonstrate that GSK Biologicals' Boostrix Polio™ vaccine is non-inferior to Sanofi-Pasteur-MSD's Tetravac™ vaccine, in terms of seroprotection rates against poliovirus type 1, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: UL of the standardised asymptotic 95% CI on the group difference [Tetravac Group minus Boostrix Polio Group] in the percentage of subjects with anti-polio type 1 antibody titers ≥ 8 was ≤ 10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.61 to 2.7]
Statistical Analysis 2: Comparison: Boostrix Polio Group vs Tetravac Group; To demonstrate that GSK Biologicals' Boostrix Polio™ vaccine is non-inferior to Sanofi-Pasteur-MSD's Tetravac™ vaccine, in terms of seroprotection rates against polio type 2, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: UL of the standardised asymptotic 95% CI on the group difference [Tetravac Group minus Boostrix Polio Group] in the percentage of subjects with anti-polio type 2 antibody titers ≥ 8 was ≤ 10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.61 to 2.7]
Statistical Analysis 3: Comparison: Boostrix Polio Group vs Tetravac Group; To demonstrate that GSK Biologicals' Boostrix Polio™ vaccine is non-inferior to Sanofi-Pasteur-MSD's Tetravac™ vaccine, in terms of seroprotection rates against polio type 3, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: UL of the standardised asymptotic 95% CI on the group difference [Tetravac Group minus Boostrix Polio Group] in the percentage of subjects with anti-polio type 3 antibody titers ≥ 8 was ≤ 10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.61 to 2.72]

4. Primary Outcome: Number of Seropositive Subjects for Anti-D and Anti-T Antibodies
Description: A seropositive subject was defined as a subject with anti-D and anti-T concentrations ≥ 0.1 IU/mL. Antibody concentrations have been assessed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 144
Participants
  Anti-D | 139 | 144
  Anti-T | 139 | 144
Statistical Analysis 1: Comparison: Boostrix Polio Group vs Tetravac Group; To demonstrate that GSK Biologicals' Boostrix Polio™ vaccine is non-inferior to Sanofi-Pasteur-MSD's Tetravac™ vaccine, in terms of seroprotection rates against diphtheria, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: Upper limit (UL) of the standardised asymptotic 95% confidence interval (CI) on the group difference [Tetravac Group minus Boostrix Polio Group] in the percentage of subjects with anti-D antibody concentrations ≥ 0.1 IU/mL was lower than or equal to (≤) 10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.61 to 2.7]
Statistical Analysis 2: Comparison: Boostrix Polio Group vs Tetravac Group; To demonstrate that GSK Biologicals' Boostrix Polio™ vaccine is non-inferior to Sanofi-Pasteur-MSD's Tetravac™ vaccine, in terms of seroprotection rates against tetanus, one month after vaccination; Test type: Non-Inferiority — Criterion for evaluation of Non-inferiority: UL of the standardised asymptotic 95% CI on the group difference [Tetravac Group minus Boostrix Polio Group] in the percentage of subjects with anti-T antibody concentrations ≥ 0.1 IU/mL was ≤ 10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-2.61 to 2.7]

5. Secondary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Antigens
Description: A seroprotected subject was defined as a subject with anti-D and anti-T concentrations ≥ 1.0 IU/mL. Antibody concentrations have been assessed by ELISA.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 144
Participants
  Anti-D | 138 | 144
  Anti-T | 137 | 143

6. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Hemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations, expressed in ELISA units per milliliter (EL.U/mL). The reference cut-off value was ≥ 5 EL.U/mL.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 144
EL.U/mL
  Anti-PT | 59.8 [52.2 to 68.5] | 75.9 [65.7 to 87.7]
  Anti-FHA | 556.2 [491.4 to 629.5] | 613.5 [547 to 688.2]
  Anti-PRN | 354.8 [280.2 to 449.4] | 7.8 [6.5 to 9.2]

7. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: A seropositive subject was defined as a subject with anti-PT, anti-FHA and anti-PRN concentrations ≥ 5.0 IU/mL. Antibody concentrations have been assessed by ELISA.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 144
Participants
  Anti-PT | 139 | 144
  Anti-FHA | 139 | 144
  Anti-PRN | 138 | 87

8. Secondary Outcome: Number of Seropositive Subjects for Anti-measles, Anti-mumps, Anti-rubella and Anti-varicella
Description: Seropositivity was defined as: subjects with antibody concentrations ≥ 150 milli-international units per milliliter (mIU/mL), ≥ 231 units per milliliter (U/mL), ≥ 4 international units per milliliter (IU/mL) and ≥ 50 mIU/mL for anti-measles, anti-mumps, anti-rubella and anti-varicella antibodies, respectively.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 146
Participants
  Anti-measles | 139 | 146
  Anti-mumps | 139 | 144
  Anti-rubella | 139 | 145
  Anti-varicella | 135 | 140

9. Secondary Outcome: Anti-measles and Anti-varicella Antibody Concentrations
Description: Antibody concentrations were assessed by ELISA, presented as geometric mean concentrations (GMCs) and expressed in mIU/mL.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 146
mIU/mL
  Anti-measles | 2743.9 [2411.4 to 3122.2] | 2863 [2534.6 to 3233.9]
  Anti-varicella | 856.7 [671.8 to 1092.4] | 909.9 [721 to 1148.2]

10. Secondary Outcome: Anti-mumps Antibody Concentrations
Description: Antibody concentrations were assessed by ELISA, presented as geometric mean concentrations (GMCs) and expressed in U/mL.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 146
U/mL | 4141.3 [3590.5 to 4776.5] | 3837.6 [3275.1 to 4496.7]

11. Secondary Outcome: Anti-rubella Antibody Concentrations
Description: Antibody concentrations were assessed by ELISA, presented as geometric mean concentrations (GMCs) and expressed in IU/mL.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 146
IU/mL | 154.5 [141.3 to 168.9] | 162.5 [145.8 to 181]

12. Secondary Outcome: Number of Subjects With Booster Responses to Anti-D and Anti-T
Description: Booster responses to anti-D and anti-T were defined as: For initially seronegative subjects (pre-vaccination concentration < cut-off of 0.1 IU/mL), antibody concentrations at least four times the assay cut-off (post-vaccination concentration ≥ 0.4 IU/mL). For initially seropositive subjects (pre-vaccination concentration ≥ 0.1 IU/mL), an increase in antibody concentrations of at least four times the pre-vaccination concentration.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 137 | 143
Participants
  Anti-D: number analyzed (Participants) | 136 | 143
  Anti-D | 130 | 136
  Anti-T | 137 | 142

13. Secondary Outcome: Number of Subjects With Booster Responses to Anti-polio Type 1, 2 and 3
Description: Booster response to the poliovirus antigens was defined as: For initially seronegative subjects (pre-vaccination antibody titre < cut-off of 8), antibody titre ≥ 32. For initially seropositive subjects (pre-vaccination antibody titres ≥ 8), an increase in antibody titres of at least four times the pre-vaccination titre.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 139 | 144
Participants
  Anti-Polio 1 | 115 | 112
  Anti-Polio 2: number analyzed (Participants) | 139 | 143
  Anti-Polio 2 | 113 | 122
  Anti-Polio 3: number analyzed (Participants) | 138 | 144
  Anti-Polio 3 | 126 | 127

14. Secondary Outcome: Number of Subjects With Booster Responses to Anti-PT, Anti-FHA and Anti-PRN
Description: Booster response to the PT, FHA and PRN antigens was defined as: For initially seronegative subjects (pre-vaccination concentration < cut-off of 5 EL.U/mL), antibody concentrations at least four times the cut-off (post-vaccination concentration ≥ 20 EL.U/mL). For initially seropositive subjects with pre-vaccination concentration ≥ 5 EL.U/mL and < 20 EL.U/mL, an increase in antibody concentrations of at least four times the pre-vaccination concentration. For initially seropositive subjects with pre-vaccination concentration ≥ 20 EL.U/mL, an increase in antibody concentrations of at least two times the pre-vaccination concentration.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 137 | 143
Participants
  Anti-PT: number analyzed (Participants) | 137 | 141
  Anti-PT | 123 | 130
  Anti-FHA: number analyzed (Participants) | 136 | 140
  Anti-FHA | 129 | 134
  Anti-PRN | 129 | 0

15. Secondary Outcome: Number of Seroconverted Subjects for Anti-measles, Anti-mumps, Anti-rubella and Anti-varicella
Description: Seroconversion for anti-measles, anti-mumps, anti-rubella and anti-varicella was defined as the appearance of antibodies after vaccination in subjects who were seronegative before vaccination. There were no seronegative subjects for anti-rubella antibodies, prior to vaccination.
Time Frame: At Month 1, one month post-vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 36 | 34
Participants
  Anti-measles: number analyzed (Participants) | 2 | 1
  Anti-measles | 2 | 1
  Anti-mumps: number analyzed (Participants) | 13 | 13
  Anti-mumps | 13 | 12
  Anti-rubella: number analyzed (Participants) | 0 | 0
  Anti-rubella | 0 | 0
  Anti-varicella | 35 | 32

16. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 151 | 152
Participants
  Any Pain | 96 | 96
  Any Redness | 58 | 66
  Any Swelling | 55 | 62

17. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache and temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 151 | 152
Participants
  Any Fatigue | 40 | 36
  Any Gastrointestinal | 23 | 15
  Any Headache | 18 | 20
  Any Temperature | 32 | 30

18. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 151 | 152
Participants | 23 | 20

19. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the whole study period (from Month 0 to Month 1)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Polio Group | Tetravac Group
Number analyzed (Participants) | 151 | 152
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Days 0-3) post-vaccination period. Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period; SAEs: during the entire study period (from Month 0 to Month 1).
Arm/Group | Boostrix Polio Group | Tetravac Group
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/152
Other Adverse Events (participants affected / at risk) | 117/151 | 117/152
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Polio Group (N=151) | Tetravac Group (N=152)
Pain (General disorders) | 96 | 96
Redness (General disorders) | 58 | 66
Swelling (General disorders) | 55 | 62
Fatigue (General disorders) | 40 | 36
Gastrointestinal (General disorders) | 23 | 15
Headache (General disorders) | 18 | 20
Temperature (General disorders) | 32 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.